CLINICAL TRIAL: NCT04261283
Title: Effects of Circuit Training on Vertigo, Oscillopsia and Dizziness in Patients With Vestibular Hypo-function
Brief Title: Circuit Training on Vertigo, Oscillopsia and Dizziness in Vestibular Hypo Function Hypo- Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/20/2001 Asna Waseem
Record Dates: First submitted 2019-12-18; First posted 2020-02-07 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Vestibular Disorder
Keywords: Dizziness; Exercise; Vestibular; Vertigo
MeSH Terms: conditions — Vestibular Diseases; Dizziness; Motor Activity; Vertigo

STUDY DESIGN:
Intervention Model Description: Two groups
Who Masked: Outcomes Assessor
Masking Description: Coding will be used and assessor will not have access to treatment allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Circuit Training (Experimental): Specific exercise are designed in circuit training
  Interventions: Other: Experimental
- Control Group (Active Comparator): Conventional treatment
  Interventions: Other: Active Comparator

INTERVENTIONS:
Other: Experimental — The Circuit Training will be consisting of:
  1. Habituation Exercises
  2. Exercises for the gaze stability (The two exercises are specifically for the patients who reported a high score on oscillopsia severity questionnaire
  3. Exercises to improve Saccade Latency.
  4. Adaptation Exercises
  5. Substitution Exercises
  6. Postural Control Exercises
  7. General Conditioning Activities
  8. Cawthorne-Cooksey Exercises
  9. Ocular Motor Exercises
  10. Gait Exercises
  11. Treatment to Decrease Sensitivity to Motion in the Environment
  Arms: Circuit Training
Other: Active Comparator — Medicines as prescribed by the ear, nose, and throat (ENT) specialist and Home-based exercise Programme (Simple and general vestibular rehabilitation exercises) will be recommended to the patients to perform. ( Not under the supervision of neuro-therapist)
  Arms: Control Group

SUMMARY:
In this research, the main purpose is to determine the effects of Circuit Training consisting of Structured Vestibular rehabilitation Program under the strict supervision of Neuro-Therapist versus Medicines and General (simple) Rehabilitation (only Home-based) in community-dwelling population of people diagnosed with Vestibular disorders. A booklet consisting of general instructions, simple vestibular exercises which are to be made a part of daily routine, specific diet plan and specific precautions to be taken by patients reporting with vertigo, oscillopsia and dizziness will also be provided to all the patients. This is a community service addition, added so that everyone in the society can have easy access to the instructions, will be cost effective, and will reduce their visits to the therapist.

DETAILED DESCRIPTION:
People diagnosed with vestibular disorders often experience dizziness , oscillopsia, trouble with vision, balance or mobility. The vestibular disorders that are called unilateral and peripheral (UPVD) are those that affect one side of the vestibular system (unilateral)and (BPVD) are those affect both sides of the vestibular system (bilateral) and only the portion of the system that is outside of the brain (peripheral-part of the inner ear). Examples of these disorders include benign paroxysmal positional vertigo (BPPV), vestibular neuritis, labyrinthitis, one-sided Ménière's disease or vestibular problems following surgical procedures such as labyrinthectomy or removal of an acoustic neuroma. Vestibular rehabilitation for these disorders is becoming increasingly used and involves various movement-based regimes.

Dizziness, oscillopsia and disequilibrium are common complaints reported by adults during visits to their doctor. Dizziness, oscillopsia, vertigo and disequilibrium are not a disease-they are symptoms that can result from a vestibular disorder or from difficulties unrelated to the inner ear, such as cardiovascular, neurological, metabolic, vision, or psychological disorders. However, as many as 45% of people with dizziness symptoms have problems in the vestibular system (balance organs of the inner ear.

Vestibular rehabilitation therapy (VRT) is an exercise-based program for reducing the symptoms of vertigo, dizziness, oscillopsia and disequilibrium with vestibular pathology (disease or disorder). A common neuro-otological approach for managing such symptoms is to prescribe medication that suppresses vestibular function. However, in the long term, such suppressants can interfere with a person's ability to make necessary adaptations. In addition, many of these medications cause drowsiness that may limit a person's ability to be active.

Vestibular habituation exercises have been recommended for these non-Ménière's patients. Although the exercises are popular, there are only a few studies in patients with chronic unilateral vestibular dysfunction. Those studies were performed with limited cases or with a wide variety of diagnoses. Herdman et al.,in their review, stressed that studies were retrospective, nonrandomized, consisting of groups that were not comparable, uncontrolled studies and, although they offer interesting descriptions of the patient population, do not provide the evidence necessary to justify the use of these exercises for treatment.

the previous study conducted a research in 2009 to find the Short-term effects of vestibular rehabilitation in patients with chronic unilateral vestibular dysfunction, a randomized controlled study. Their objective was to evaluate the short-term effects of vestibular rehabilitation on a symptom, disability, balance, and postural stability in patients with chronic unilateral vestibular dysfunction. Significant improvements were seen in symptom, disability, balance, and postural stability in chronic unilateral vestibular dysfunction after an exercise program.

in 2013 study was conducted on finding out the effects of Vestibular rehabilitation with virtual reality in Meniere disease. Their aim was to verify the effect of a virtual reality-based balance rehabilitation program for patients with Meniere disease. They concluded that Virtual reality-based balance rehabilitation effectively improved dizziness, quality of life, and limit of stability of patients with Meniere's disease.

in 2006 a study was conducted to Compare between Oculomotor Rehabilitation and Vestibular Electrical Stimulation in Unilateral Peripheral Vestibular Deficit. The aim of their study was to evaluate the effects of oculomotor rehabilitation (group 2) on static balance and a dizziness handicap and to compare those with the effects to vestibular electrical stimulation (group 1). Analysis of the equilibrium system subcomponents did not show any variation. Oculomotor exercises, employed in most rehabilitative protocols and including head movements to improve vestibular adaptation, have proved to reduce the perceived overall impairment and postural sway in patients with recent unilateral vestibular disorders, even though the disorders are not associated with head movements. Comparison of our two study groups did not show any significant difference, revealing that both forms of therapy are effective.

in 2013, a study evaluated the feasibility of integrating vestibular rehabilitation and cognitive behaviour therapy (VR-CBT) for people with persistent dizziness in primary care. This was a prospective single-group pre- and post-test study. Participants reported that the VR-CBT was relevant and led to an improvement in function.Dizziness Handicap Inventory (DHI) scores improved beyond a minimal important change in two out of five participants, and preferred gait velocity increased beyond a minimal important change in two out of three participants. The current tests and VR-CBT treatment protocols were feasible. Some changes are suggested to optimize the protocols, before conducting a randomized controlled trial.

Up-till now a properly structured Circuit Training consisting of Vestibular Rehabilitation exercises, in which each exercise is designed such that it specifically focus on each and every symptom separately has not developed. So, in this research a Circuit Training consisting of Vestibular exercises, each exercise included is focusing on a specific goal separately

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with Vestibular Disorders/
* patient with Dysfunctions by ENT specialist.

Exclusion Criteria:

Patients diagnosed with BPPV.

* Central nervous system (CNS) involvement (significant neurological disorders)
* Musculoskeletal (MSK) system deficits (orthopedic disorders)
* Uncontrolled hypertension (HTN)
* Heart diseases
* Psychosocial abnormalities
* Psychiatric disorders

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Visual Vertigo Analogue Scale | 4 week
  changes from the baseline,this scale is used to measure the intensity of symptoms, 0-10 cm line zero anchor representing no dizziness and 10 anchor representing extreme dizziness or activity avoided due to dizziness
Vertigo Handicap Questionnaire | 4 week
  changes from the baseline, this scale is used to assess the disability level in vestibular impairment. 25 Items measuring Four dimensions(restriction of Activity, social Anxieties, fear of Vertigo, severity of episodes). Item scaling is on 5 points likert scale from 0 (no handicap) to 4 (maximum handicap)
Dizziness Handicap Inventory | 4 week
  changes from the baseline, this test is used to determine the physical, functional and emotional components of Dizziness. Item Scores are summed, there is a maximum score of 100 (28 points for physical, 36 for emotional and 36 for functional and a minimum score of 0. The higher the score, the greater the perceived handicap due to dizziness. Answers are graded: 0 (no), 2 (sometimes), 4 (Yes)

SECONDARY OUTCOMES:
Vestibular Disorders Activities of Daily Living Scale | 4 week
  changes from the baseline , this is scale used to asses the level of activities
Berg Balance Scale | 4 week
  changes from the baseline, Berg balance scale is used for functional balance. participants are asked to perform 14 tasks frequently used in daily life activities. The highest possible score is 56 points. A higher score indicates better balance.

CONTACTS AND LOCATIONS:
Overall Officials: Arshad Nawaz AN Malik, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Later on will be publish

REFERENCES:
- [Background] Johansson M, Akerlund D, Larsen HC, Andersson G. Randomized controlled trial of vestibular rehabilitation combined with cognitive-behavioral therapy for dizziness in older people. Otolaryngol Head Neck Surg. 2001 Sep;125(3):151-6. doi: 10.1067/mhn.2001.118127. PMID 11555746
- [Background] Herdman SJ, Blatt PJ, Schubert MC. Vestibular rehabilitation of patients with vestibular hypofunction or with benign paroxysmal positional vertigo. Curr Opin Neurol. 2000 Feb;13(1):39-43. doi: 10.1097/00019052-200002000-00008. PMID 10719648
- [Background] Giray M, Kirazli Y, Karapolat H, Celebisoy N, Bilgen C, Kirazli T. Short-term effects of vestibular rehabilitation in patients with chronic unilateral vestibular dysfunction: a randomized controlled study. Arch Phys Med Rehabil. 2009 Aug;90(8):1325-31. doi: 10.1016/j.apmr.2009.01.032. PMID 19651266
- [Background] Kristiansen L, Magnussen LH, Juul-Kristensen B, Maeland S, Nordahl SHG, Hovland A, Sjobo T, Wilhelmsen KT. Feasibility of integrating vestibular rehabilitation and cognitive behaviour therapy for people with persistent dizziness. Pilot Feasibility Stud. 2019 May 20;5:69. doi: 10.1186/s40814-019-0452-3. eCollection 2019. PMID 31139431